CLINICAL TRIAL: NCT07077122
Title: Evaluation of the Systemic Burden of Non-surgical Periodontal Therapy: A Randomized Clinical Trial on Five Different Treatment Protocols
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Evangelia Zampa, Principal investigator - DDS, MSc, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 688/11.02.2025; Ethics committee (Other: Dental School of Athens, NKUA)
Record Dates: First submitted 2025-06-30; First posted 2025-07-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis
Keywords: periodontitis; inflammatory markers; non-surgical periodontal therapy; bacteremia
MeSH Terms: conditions — Periodontitis; Bacteremia | interventions — Tooth Exfoliation; Root Planing; Antibiotic Prophylaxis; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Full-Mouth SRP (Experimental): oral hygiene instructions and full mouth scaling and root planing in 24 hours. Clinical re-evaluation in 8 weeks.
  Interventions: Procedure: Scaling and Root Planing
- SRP + Antibiotics (Experimental): oral hygiene instructions and full mouth scaling and root planing in 24 hours along with antibiotic prophylaxis. Clinical re-evaluation in 8 weeks.
  Interventions: Procedure: Scaling and Root Planing; Drug: antibiotic prophylaxis
- SRP + Laser (Experimental): oral hygiene instructions and 810nm diode laser at the base of the gingival sulcus/pocket following by full mouth scaling and root planing in 24 hours. Clinical re-evaluation in 8 weeks.
  Interventions: Procedure: Scaling and Root Planing; Device: 810nm Diode Laser
- SRP + Air Polishing (Experimental): oral hygiene instructions and air polishing following by full mouth scaling and root planing in 24 hours. Clinical re-evaluation in 8 weeks.
  Interventions: Procedure: Scaling and Root Planing; Procedure: Air Polishing
- Quadrant SRP (Control) (Active Comparator): Oral hygiene instructions, scaling and root planing per quadrant with an interval of 7 days per session. Clinical re-evaluation in 8 weeks after last session.
  Interventions: Procedure: Scaling and Root Planing

INTERVENTIONS:
Procedure: Scaling and Root Planing — Mechanical debridement of tooth surfaces using hand and ultrasonic instruments
Drug: antibiotic prophylaxis — 2g Amoxicillin given 1 hour prior to instrumentation
  Arms: SRP + Antibiotics
Device: 810nm Diode Laser — Laser applied at base of gingival pockets prior to mechanical debridement.
  Arms: SRP + Laser
Procedure: Air Polishing — air flow-based mechanical debridement with erythritol powder
  Arms: SRP + Air Polishing

SUMMARY:
Periodontitis is a chronic inflammatory disease of the periodontal tissues leading to the destruction of the tooth supporting structures. Despite the fact that periodontal bacteria are etiological agents, host susceptibility related to the inflammatory response to plaque bacteria is the main determinant of the development of periodontitis. Non-surgical periodontal therapy (NSPT) represents the base of any therapeutic approach. Its main component is the removal of bacterial deposits, i.e. soft biofilm or mineralized calculus, from the tooth surface via mechanical debridement.

It is well established that patients suffering from periodontitis present with a low-grade systemic inflammatory state when compared to healthy subjects. Increased concentrations of inflammatory biomarkers in systemic circulation, such as, C-reactive protein (CRP) and interleukin (IL)-6, have already been reported. A significant amount of evidence derived from epidemiological as well as experimental studies has implicated periodontitis as a putative risk factor for a number of systemic diseases, such as, cardiovascular diseases, diabetes and respiratory diseases having systemic low-grade inflammation as their underlying pathogenic mechanism. Furthermore, several intervention studies provide evidence that periodontal treatment may improve systemic inflammatory markers and potentially reduce the risk for cardio-metabolic diseases.

However, periodontal therapy may pose a transient, short-term health hazard immediately after instrumentation of the root surface presumably due to the spill of bacteria and their products in the systemic circulation and the subsequent acute inflammatory response. Positive bacteremia in NSPT ranges from 13% to 80.9% after mechanical debridement depending primarily on the periodontal status of the patient, but also on the study design and the microbiological methodology.

Finally, an important aspect concerning NSPT is method and duration of delivery. NSPT may be carried out with either hand instruments, power driven instruments, such as, ultrasonic and sonic or a "blended approach" using both. Besides these instruments, the adjunctive use of lasers or/and air powder technology has been proposed. Regarding duration, treatment may be staged over several visits with a quadrant approach, or with a full-mouth debridement approach, also referred to as an intensive treatment approach, which delivers complete debridement within 24 hours.

The aim of this clinical trial is to assess the immediate systemic burden of five different treatment protocols for the NSPT on:

1. bacteremia
2. serum inflammatory responses. Additionally, saliva CRP levels will be assessed and compared to serum. Moreover, the effectiveness of the treatment protocols on clinical periodontal parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis stage III or IV
* Non-smokers or light smokers (<10 cigarettes/day)
* No NSAIDs in regular basis or antibiotics 3 months before
* No previous periodontal treatment 12 months before
* No presence of other acute or chronic infections
* No systemic disease or medication known to affect the serum level of inflammatory markers (cyclooxygenase inhibitors, platelet aggregation inhibitors, lipid lowering agents, â-adrenoreceptor antagonists, angiotensin converting enzyme inhibitors, antidiabetic agents, estrogen-based medications, medication for autoimmune disease, magnesium or vitamin E supplements)
* No pregnancy or lactation
* Written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in serum high-sensitivity C-reactive protein (hs-CRP) levels | Baseline-7 days after the last periodontal session
  For hs-CRP, blood would be collected:
  * Before each periodontal session
  * 24 hours after each periodontal session
  * 7 days after each periodontal session

SECONDARY OUTCOMES:
Changes in serum Interleukin 6 (IL-6) | Baseline-7 days after the last periodontal session
  For IL-6, blood would be collected:
  * Before each periodontal session
  * 24 hours after each periodontal session
  * 7 days after each periodontal session
Presence and load of bacteremia | Baseline-15 minutes after the last periodontal session
  culture, PCR, 16S rRNA sequencing
Changes in mean Clinical Attachment Level (CAL) | Baseline-8 weeks after the last periodontal session
  CAL would be assessed before treatment initiation and would then be recorded at 8 weeks after the last periodontal session.
  All clinical measurements would be taken using a manual probe. CAL would be recorded at six sites per tooth. Third molars would be excluded from the measurements.
Salivary CRP correlation with serum CRP | Baseline-7 days after the last periodontal session
  saliva CRP levels will be assessed and compared to serum
Changes in serum Tumor Necrosis Factor a (TNF-a) levels | Baseline-7 days after the last periodontal session
  For changes in TNF-a levels, blood would be collected:
  * Before each periodontal session
  * 24 hours after each periodontal session
  * 7 days after each periodontal session
Changes in Serum amyloid A (SAA) levels | Baseline-7 days after the last periodontal session
  For changes in SAA levels, blood would be collected:
  * Before each periodontal session
  * 24 hours after each periodontal session
  * 7 days after each periodontal session
Changes in Serum cystatin c levels | Baseline-7 days after the last periodontal session
  For changes in serum cystatin c levels, blood would be collected:
  * Before each periodontal session
  * 24 hours after each periodontal session
  * 7 days after each periodontal session
Changes in Matrix metalloproteinase-8 (MMP-8) levels | Baseline-7 days after the last periodontal session
  For changes in MMP-8 levels, blood would be collected:
  * Before each periodontal session
  * 24 hours after each periodontal session
  * 7 days after each periodontal session
Changes in serum D-dimers levels | Baseline-7 days after the last periodontal session
  For changes in serum D-dimers levels, blood would be collected:
  * Before each periodontal session
  * 24 hours after each periodontal session
  * 7 days after each periodontal session
Changes in serum Lipopolysaccharide (LPS) levels | Baseline-7 days after the last periodontal session
  For changes in serum LPS levels, blood would be collected:
  * Before each periodontal session
  * 24 hours after each periodontal session
  * 7 days after each periodontal session
Changes in mean Pocket Depth (PD) | Baseline-8 weeks after the last periodontal session
  PD would be assessed before treatment initiation and would then be recorded at 8 weeks after the last periodontal session.
  All clinical measurements would be taken using a manual probe. PD would be recorded at six sites per tooth. Third molars would be excluded from the measurements.
Changes in mean Gingival Recession (GR) | Baseline-8 weeks after the last periodontal session
  GR would be assessed before treatment initiation and would then be recorded at 8 weeks after the last periodontal session.
  All clinical measurements would be taken using a manual probe. GR would be recorded at six sites per tooth. Third molars would be excluded from the measurements.
Changes in Full-Mouth Plaque Score (FMPS) | Baseline-8 weeks after the last periodontal session
  FMPS would be assessed before treatment initiation and would then be recorded at 8 weeks after the last periodontal session.
  All clinical measurements would be taken using a manual probe. FMPS would be recorded at six sites per tooth. Third molars would be excluded from the measurements.
Changes in Full-Mouth Bleeding Score (FMBS) | Baseline-8 weeks after the last periodontal session
  FMBS would be assessed before treatment initiation and would then be recorded at 8 weeks after the last periodontal session. All clinical measurements would be taken using a manual probe. FMBS would be recorded at six sites per tooth. Third molars would be excluded from the measurements.
Changes in simplified gingival index (s-GI) | Baseline-8 weeks after the last periodontal session
  s-GI would be assessed before treatment initiation and would then be recorded at 8 weeks after the last periodontal session. All clinical measurements would be taken using a manual probe. s-GI would be recorded at four sites per tooth. Third molars would be excluded from the measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Madianos Phoebus, Study Chair — Professor
Locations (1):
- Department of Periodontology, Dental School of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Time Frame: After publication of the main study results.
Access Criteria: Data will be available upon reasonable request to qualified researchers for academic purposes.

REFERENCES:
- [Background] Sanz M, Marco Del Castillo A, Jepsen S, Gonzalez-Juanatey JR, D'Aiuto F, Bouchard P, Chapple I, Dietrich T, Gotsman I, Graziani F, Herrera D, Loos B, Madianos P, Michel JB, Perel P, Pieske B, Shapira L, Shechter M, Tonetti M, Vlachopoulos C, Wimmer G. Periodontitis and cardiovascular diseases: Consensus report. J Clin Periodontol. 2020 Mar;47(3):268-288. doi: 10.1111/jcpe.13189. Epub 2020 Feb 3. PMID 32011025
- [Background] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Background] Kinane DF, Riggio MP, Walker KF, MacKenzie D, Shearer B. Bacteraemia following periodontal procedures. J Clin Periodontol. 2005 Jul;32(7):708-13. doi: 10.1111/j.1600-051X.2005.00741.x. PMID 15966875